CLINICAL TRIAL: NCT06293235
Title: Investigating Male Factors and Their Relationships With Reproductive Health Outcomes in Singapore: Towards Optimal Fertility, Fathering and Fatherhood studY
Brief Title: Towards Optimal Fertility, Fathering and Fatherhood studY
Acronym: TOFFFY
Status: Recruiting | Type: Observational
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2024/2120
Record Dates: First submitted 2024-02-20; First posted 2024-03-05 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-02

CONDITIONS: Reproductive Issues; Fertility Issues
Keywords: Male; Risk factor; Lifestyle; Semen analysis; Epigenetic; Oxidative stress; DNA fragmentation
MeSH Terms: conditions — Infertility | interventions — Semen Analysis; Amino Acid Motifs

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subfertile couples: Couples who are not able to conceive for at least 12 months with female partners without infertility diagnosis.
  Interventions: Other: Lifestyle and metabolic indicators
- Fertile couples: Couples with attempted time to conceive within 12 months to achieve this pregnancy or with unplanned pregnancy, with female partners who are currently pregnant with viable intrauterine pregnancy.
  Interventions: Other: Lifestyle and metabolic indicators

INTERVENTIONS:
Other: Lifestyle and metabolic indicators — Socio-demographics, health history, behavioural characteristics, environmental exposures, anthropometric measurements, body fat composition, metabolic and stress biomarkers, semen physical and molecular characteristics.
  Other Names: Semen quality and characteristics

SUMMARY:
This case-control study involving fertile and subfertile couples aims to identify male factors related to pregnancy likelihood, create a fertility index measure combining male and female factors to predict pregnancy likelihood, and examine how male factors relate to the semen physical and biological characteristics.

DETAILED DESCRIPTION:
Paternal contributions to fertility and reproductive health outcomes have been understudied, despite promising evidence from animal studies. This study aims to investigate the male contribution to pregnancy likelihood and explore the underlying biological mechanisms. Specifically, the investigators aim to (1) identify male factors associated with pregnancy rate; (2) develop a fertility index combining modifiable factors for both males and females to predict pregnancy rate; and (3) explore the relationship of male modifiable factors with semen physical and molecular characteristics. This is a case-control study with 480 fertile and subfertile males (along with their female partners), recruited from KK Women's and Children's Hospital. The investigators will use questionnaires to collect data on socio-demographic characteristics, clinical, lifestyle, and environmental factors; analyze metabolic and stress biomarkers from blood samples; and measure semen parameters including sperm motility, density, morphology, volume, DNA fragmentation, DNA methylation, gene expression, and seminal plasma oxidative status. Findings from this proposed study will pave the way for developing lifestyle-based or medical interventions to enhance male and couple reproductive health, and potentially benefiting future offspring health.

ELIGIBILITY:
Inclusion Criteria:

Subfertile couples:

* men aged ≥21-49 years
* men with a female partner aged 21-39 years
* couples who are not able to conceive for at least 12 months
* couples who are Singapore citizen or permanent resident

Fertile couples:

* men aged 21-49 years
* men with a female partner aged 21-39 years
* men with proven fertility defined as those female partners who are currently pregnant and with viable intrauterine pregnancy at gestational weeks of less or equal to 16 at the time of the study
* couples with attempted time to conceive within 12 months to achieve this pregnancy or with unplanned pregnancy
* couples who are Singapore citizen or permanent resident

Exclusion Criteria:

Subfertile couples:

* male infertility of a known aetiology including azoospermia, retrograde ejaculation, genetic disorders, cancer treatment, or testes trauma
* female infertility diagnosis as confirmed by diagnostic imaging or having severe endometriosis
* female partners with irregular menstrual cycle >35 days
* couples with known chromosomal abnormalities

Fertile couples:

* couples who achieve pregnancy after oocyte or spermatozoa donation
* couples with known chromosomal abnormalities
* female partners with known uterine abnormalities

Ages: 21 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Based on biological sex identity for males and females
Study Population: The subfertile couples will be recruited from the infertility clinics, while the fertile couples will be recruited from the antenatal clinics. Both groups will also be recruited from on-going preconception and pregnancy programs in the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 960 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rate | Up to 16 weeks of gestation
  Defined by viable intrauterine pregnancy at gestational weeks of less or equal to 16 at the time of the study

SECONDARY OUTCOMES:
Fertility index | Through study completion, an average of 3 years
  Defined by a composite index score derived from both male and female predictive factors
Oxidative stress | Through study completion, an average of 3 years
  Defined by oxidative status measured from blood and semen samples using the micro-NMR
Semen volume | Up to 2 years
  Assessed by semen analysis in ml
Sperm concentration | Up to 2 years
  Assessed by semen analysis in million/ml
Sperm total motility | Up to 2 years
  Assessed by semen analysis in percent
Sperm progressive motility | Up to 2 years
  Assessed by semen analysis in percent
Total progressive motile sperm count | Up to 2 years
  measured by multiplying the semen volume (ml) by sperm concentration (million/ml) and the percentage of progressively motile sperm
Single strand sperm DNA fragmentation | Up to 2 years
  Measured by the AI-powered semen analyzer
Double strand sperm DNA fragmentation | Up to 2 years
  Measured by the AI-powered semen analyzer
mRNA level | Through study completion, an average of 3 years
  From blood and semen samples through transcriptomics analysis
sncRNA level | Through study completion, an average of 3 years
  From blood and semen samples through transcriptomics analysis
DNA methylation | Through study completion, an average of 3 years
  From blood and semen samples through bisulfite sequencing

OTHER OUTCOMES:
Sperm morphology | Up to 2 years
  Assessed by semen analysis

CONTACTS AND LOCATIONS:
Overall Officials: See Ling Loy, PhD, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ku CW, Pek JW, Cheung YB, Tharmalingam Durgahshree MD, Chan M, Lee YH, Godfrey K, Yap F, Chan JKY, Loy SL. Investigating male factors and their relationships with reproductive health outcomes: a case-control study protocol for Towards Optimal Fertility, Fathering, and Fatherhood studY (TOFFFY) in Singapore. BMJ Open. 2025 Jan 15;15(1):e088143. doi: 10.1136/bmjopen-2024-088143. PMID 39819913